CLINICAL TRIAL: NCT06681480
Title: Transcranial Magnetic Stimulation (rTMS) for the Treatment of Focal Refractory Epilepsy: Neuropsychological and Electrophysiological Evaluation.
Brief Title: Transcranial Magnetic Stimulation (rTMS) for Refractory Focal Epilepsy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Comenius University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: U-1111-1280-4605; UK/33/2022 (Other Grant/Funding Number: Comenius University)
Record Dates: First submitted 2022-09-09; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Focal Epilepsy; Transcranial Magnetis Stimulation
Keywords: Epilepsy, Focal, Partial, Central Nervous System Diseases, Brain Diseases
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy; Central Nervous System Diseases; Brain Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention/treatment (Experimental): figure-of-eight active rTMS coil rTMS is administered using the figure-of-eight active coil, at 90% of the resting motor threshold over the epileptogenic region, in trains with a total of 15000 pulses during 5 weekdays at low frequency 0,5Hz Device: figure-of-eight active rTMS coil navigated rTMS over epileptogenic focus using figure-of-eight active rTMS coil, optic navigation system
  Interventions: Device: figure-of-eight active rTMS coil device
- Control arm (Sham Comparator): figure-of-eight active rTMS coil rTMS is administered using the figure-of-eight sham coil, at 90% of the resting motor threshold over the epileptogenic region, in trains with a total of 15000 pulses during 5 weekdays at sham stimulation Device: figure-of-eight sham rTMS coil navigated rTMS over epileptogenic focus using figure-of-eight sham rTMS coil, optic navigation system
  Interventions: Device: figure-of-eight sham rTMS coil device

INTERVENTIONS:
Device: figure-of-eight active rTMS coil device — rTMS is administered using the figure-of-eight active coil, at 90% of the resting motor threshold over the epileptogenic region, in trains with a total of 15000 pulses during 5 weekdays at low frequency 0,5Hz Device: figure-of-eight active rTMS coil navigated rTMS over epileptogenic focus using figure-of-eight active rTMS coil, optic navigation system
  Arms: Intervention/treatment
Device: figure-of-eight sham rTMS coil device — rTMS is administered using the figure-of-eight sham coil, in trains with a total of 15000 pulses during 5 weekdays Device: figure-of-eight sham rTMS coil navigated rTMS over epileptogenic focus using figure-of-eight sham rTMS coil, optic navigation system
  Arms: Control arm

SUMMARY:
Epilepsy as a brain disease is characterised by enhanced brain excitability. Low frequency repetitive transcranial magnetic stimulation (rTMS) can be an effective treatment for refractory focal epilepsy. Today different ways of stimulation were used, the best protocol of rTMS in refractory focal epilepsy is under evaluation. The aim of our study is neuropsychological and electrophysiological evaluation before and after rTMS sessions, the results of rTMS will be compared with VNS outcome in patients, who undergoes VNS implantation after rTMS.

DETAILED DESCRIPTION:
1. Background Epilepsy is a chronic disease that causes repetitive seizures. In 60% to 70% of people with epilepsy (PWE) , these seizures start in a small part of the brain (focal epilepsy). Up to 30% of people with epilepsy continue to have seizures despite optimal pharmacological care. Invasive methods - called epilepsy surgery are the choice of treatment for this group of the patients. New non- invasive non- pharmacological methods are on the way.
2. Aim of the study Treatment the people with focal epilepsy with non- invasive transcranial magnetic stimulation (rTMS) to the region that causes the epilepsy. A part of the patients will after that be treated with invasive VNS implantation. The aim is to evaluate neuropsychological and electrophysiological out come in non- invasive arm and in combined arm (VNS after rTMS).
3. Inclusion criteria The patients with neocortical focal epilepsy older than 18 years, not controlled with antiseizure drugs, with confirmed refractory epilepsy.
4. Study methodology The seizure frequency will be controlled with seizure diaries, patients will be evaluated in tertiary epilepsy centre. The patients will be on stable dose of drugs 4 week before and at least 8 weeks after last TMS session. They will be evaluated by battery of neuropsychological tests (cognition, emotions, personality) and electrophysiological methods ( QEEG, SEP n. medianus) before rTMS sessions and after rTMS session and a month later. A part of the patient, who will continue to VNS implantation will be evaluated before VNS implantation and 6 month later again.

   The magnetic pulses will be delivered in a active session or in a placebo session ( sham). The investigators will not tell in which order they deliver the treatments.
5. What are the possible benefits and risks of participating? The investigators believe, that the patients will have fewer seizures in the weeks following the active treatment and that the improvement could be detected in neuropsychological evaluations and in electrophysiology. It is not known, if the results of rTMS could predict the response of the patients to VNS stimulation.

ELIGIBILITY:
Inclusion Criteria:

- fully characterized refractory focal neocortical epilepsy (i.e. the epileptogenic zone is well defined) on a stable drug regimen for at least one month, able to complete a seizure dairy either by the patient or by a significant other

Exclusion Criteria:

- Metal in the head including deep brain stimulators, aneurysmal clips, ventricular shunts, cochlear implants, ossicular reconstruction of the middle ear, VNS implants pacemaker, implantable cardioverter-defibrillator (ICD) psychogenic non-epileptic seizures and other non-epileptic spells

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Seizure frequency and severity | 1 hour
  50% Responder Rate after active rTMS treatment and median of seizure frequency reduction from baseline according seizure diaries of the patients rated per 28 day period

SECONDARY OUTCOMES:
QOLIE-31-P measurement of different neuropsychological aspects of epilepsy | 20 min
  measurement of different neuropsychological aspects of epilepsy (cognition, emotions, social well- being and social functioning) in patients before and one month after rTMS: Questionnaires: Quality of Life in Epilepsy- problems (QOLIE-31-P) change of score
Electrophysiological evaluation with quantitative EEG | 30 min
  Electrophysiological evaluation with quantitative EEG ( QEEG) as response to rTMS stimulation and correlation with primary outcome measure and neuropsychological outcome measured with neuropsychological batteries change in cordance
Comparison the data in the group of the patients | 1 hour
  Comparison the data in the group of the patients, who will after rTMS continue to VNS implantation, multiregression analysis for possible connection between rTMS response and later VNS efficacy
Drop out rate and adverse event profile | 1 hour
  Drop out rate and adverse event profile
LSSS- measurement of different neuropsychological aspects of epilepsy | 10 min
  measurement of different neuropsychological aspects of epilepsy (cognition, emotions, social well- being and social functioning) in patients before and one month after rTMS: Liverpool seizure severity scale (LSSS) change in frequency and severity of seizures
PHQ-9 measurement of different neuropsychological aspects of epilepsy | 5 min
  measurement of different neuropsychological aspects of epilepsy (cognition, emotions, social well- being and social functioning) in patients before and one month after rTMS: Patients Health Questionnaire ( PHQ-9), change of score
GAD-7 measurement of different neuropsychological aspects of epilepsy | 5 min
  measurement of different neuropsychological aspects of epilepsy (cognition, emotions, social well- being and social functioning) in patients before and one month after rTMS: Generalized Anxiety Disorder(GAD-7), change of score
ROCFT measurement of different neuropsychological aspects of epilepsy | 10 min
  measurement of different neuropsychological aspects of epilepsy (cognition, emotions, social well- being and social functioning) in patients before and one month after rTMS: Rey-Osterrieth complex figure test ( ROCFT), change of score
STROOP measurement of different neuropsychological aspects of epilepsy | 15 min
  measurement of different neuropsychological aspects of epilepsy (cognition, emotions, social well- being and social functioning) in patients before and one month after rTMS: Stroop 1,2,3, change of score
TMT AB measurement of different neuropsychological aspects of epilepsy | 5 min
  measurement of different neuropsychological aspects of epilepsy (cognition, emotions, social well- being and social functioning) in patients before and one month after rTMS: Trail making test A,B, (TMT AB), change of score
DST measurement of different neuropsychological aspects of epilepsy | 10 min
  measurement of different neuropsychological aspects of epilepsy (cognition, emotions, social well- being and social functioning) in patients before and one month after rTMS: Digit span test (DST), change of score
AVLT measurement of different neuropsychological aspects of epilepsy | 10 min
  measurement of different neuropsychological aspects of epilepsy (cognition, emotions, social well- being and social functioning) in patients before and one month after rTMS: Auditory verbal learning test ( AVLT), change of score
MoCA measurement of different neuropsychological aspects of epilepsy | 20 min
  measurement of different neuropsychological aspects of epilepsy (cognition, emotions, social well- being and social functioning) in patients before and one month after rTMS: Montreal Cognitive Assessment (MoCA) change of score
SDMT measurement of different neuropsychological aspects of epilepsy | 10 min
  measurement of different neuropsychological aspects of epilepsy (cognition, emotions, social well- being and social functioning) in patients before and one month after rTMS: Symbol Digit Modalities Test (SDMT), change of score
StT measurement of different neuropsychological aspects of epilepsy | 10 min
  measurement of different neuropsychological aspects of epilepsy (cognition, emotions, social well- being and social functioning) in patients before and one month after rTMS: Story Test (StT), change of score
WCST measurement of different neuropsychological aspects of epilepsy | 10 min
  measurement of different neuropsychological aspects of epilepsy (cognition, emotions, social well- being and social functioning) in patients before and one month after rTMS: Wisconsin Card Sorting Test (WCST), change of score
Electrophysiological evaluation with quantitative SEP | 1 hour
  Electrophysiological evaluation with SEP (n. medianus amplitude) as response to rTMS stimulation and correlation with primary outcome measure and neuropsychological outcome measured with neuropsychological batteries change of amplitude

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Department of Neurology, Faculty of Medicine COMENIUS UNIVERSITY BRATISLAVA, Bratislava, Slovak Republic, Slovakia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sun W, Mao W, Meng X, Wang D, Qiao L, Tao W, Li L, Jia X, Han C, Fu M, Tong X, Wu X, Wang Y. Low-frequency repetitive transcranial magnetic stimulation for the treatment of refractory partial epilepsy: a controlled clinical study. Epilepsia. 2012 Oct;53(10):1782-9. doi: 10.1111/j.1528-1167.2012.03626.x. Epub 2012 Sep 5. PMID 22950513
- [Background] Fregni F, Otachi PT, Do Valle A, Boggio PS, Thut G, Rigonatti SP, Pascual-Leone A, Valente KD. A randomized clinical trial of repetitive transcranial magnetic stimulation in patients with refractory epilepsy. Ann Neurol. 2006 Oct;60(4):447-55. doi: 10.1002/ana.20950. PMID 17068786
- [Background] Pereira LS, Muller VT, da Mota Gomes M, Rotenberg A, Fregni F. Safety of repetitive transcranial magnetic stimulation in patients with epilepsy: A systematic review. Epilepsy Behav. 2016 Apr;57(Pt A):167-176. doi: 10.1016/j.yebeh.2016.01.015. Epub 2016 Mar 10. PMID 26970993
- [Background] Seynaeve L, Devroye A, Dupont P, Van Paesschen W. Randomized crossover sham-controlled clinical trial of targeted low-frequency transcranial magnetic stimulation comparing a figure-8 and a round coil to treat refractory neocortical epilepsy. Epilepsia. 2016 Jan;57(1):141-50. doi: 10.1111/epi.13247. Epub 2015 Dec 8. PMID 26642974
- [Background] Cantello R, Rossi S, Varrasi C, Ulivelli M, Civardi C, Bartalini S, Vatti G, Cincotta M, Borgheresi A, Zaccara G, Quartarone A, Crupi D, Lagana A, Inghilleri M, Giallonardo AT, Berardelli A, Pacifici L, Ferreri F, Tombini M, Gilio F, Quarato P, Conte A, Manganotti P, Bongiovanni LG, Monaco F, Ferrante D, Rossini PM. Slow repetitive TMS for drug-resistant epilepsy: clinical and EEG findings of a placebo-controlled trial. Epilepsia. 2007 Feb;48(2):366-74. doi: 10.1111/j.1528-1167.2006.00938.x. PMID 17295632
- [Derived] Melus J, Waczulikova I, Hapakova L, Konecna M, Valkovic P, Timarova G. Repetitive transcranial magnetic stimulation for the treatment of focal drug-resistant epilepsy: A crossover, randomized, single-blinded, sham-controlled clinical trial. Seizure. 2025 Sep;131:290-297. doi: 10.1016/j.seizure.2025.07.015. Epub 2025 Jul 27. PMID 40782718